CLINICAL TRIAL: NCT00354887
Title: A Phase II Study of Capecitabine and Oxaliplatin (XELOX) in Adenocarcinoma of the Small Bowel and Ampulla of Vater
Brief Title: Capecitabine and Oxaliplatin in Adenocarcinoma of the Small Bowel and Ampulla of Vater
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0827
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Results first posted 2011-07-14 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastrointestinal Cancer; Small Bowel Cancer; Ampulla of Vater; Capecitabine; Xeloda; Oxaliplatin; Eloxatin
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin + Capecitabine (Experimental): Intravenous Oxaliplatin 130 mg/m^2, Day 1 + Oral Capecitabine 750 mg/m^2 twice daily Days 1-14.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — Oral capecitabine 750 mg/m^2 twice daily (total daily dose 1500 mg/m^2) on Days 1-14 in 21 Day Cycle.
  Other Names: Xeloda
Drug: Oxaliplatin — 130 mg/m^2 by vein Day 1 over 2 hours in 21 Day Cycle
  Other Names: Eloxatin

SUMMARY:
Primary Objective:

1. To determine the objective response rate (complete plus partial) to the combination of capecitabine (Xeloda) and oxaliplatin (Eloxatin) (XELOX) in patients with adenocarcinoma of the small bowel and ampulla of Vater.

Secondary objectives include determining the toxicity, time-to-treatment failure, and overall survival rates in patients treated with this combination.

DETAILED DESCRIPTION:
Oxaliplatin is a chemotherapy drug designed to destroy cancer cells by interfering with DNA function, which is necessary for growth of new cells.

Capecitabine is a chemotherapy drug designed to destroy cancer cells by interfering with cell division, which is important to the growth of cancer.

You will receive 14 days of treatment followed by 7 days without treatment, 21 days in all, otherwise known as a "cycle" of therapy. On Day 1 of each cycle, you will receive oxaliplatin injected into a vein over a period of 2 hours. For this injection, you will need to have a small tube inserted into a vein under the skin of the chest (central venous line) to receive oxaliplatin. Oxaliplatin must be given at M.D. Anderson.

You will take capecitabine tablets twice a day for the first two weeks (Days 1-14) of each 3-week cycle. No treatment will be given for the next 7 days. You must take capecitabine within 30 minutes after breakfast and dinner, with morning and evening doses about 12 hours apart. You should take capecitabine by mouth with water, and not fruit juices. At the first treatment visit and every 3 weeks, you will receive enough capecitabine to last until the next visit. At each visit, you must return any capecitabine you have not used as well as all empty bottles.

During Cycle 1, routine blood tests (about 2 teaspoons of blood) will be done once a week. Before each new cycle of therapy, you will have a complete physical exam and blood (about 2 ½ teaspoons) will be collected for routine tests. You will be asked by the study doctor about all medications you have taken since starting the study drugs and any health problems that you may have experienced. Also, you will have an x-ray or computed tomography (CT) scan of the chest and either CT scans or magnetic resonance imaging (MRIs) of the tumor(s) every 3 cycles and at the end of the study. Additional tests may be done during the study if your doctor feels it is necessary for your care.

This study will require you to receive at least 3 cycles of treatment. However, if you experience severe side effects or your disease becomes worse, treatment may be delayed, stopped, or you may receive smaller doses of the treatment. You may continue to receive treatment on this study until the disease gets worse or you experience any intolerable side effects. If this happens, you will be taken off the study and your doctor will discuss other treatment options with you.

When you stop taking part in the study, you will have blood (about 3 teaspoons) collected for routine tests. You will have a physical exam and either a CT scan or an MRI to check on the status of the disease. You will be contacted by phone every three months for the rest of your life to check on your state of health and ask you about further symptoms you may be experiencing.

This is an investigational study. The drugs oxaliplatin and capecitabine are FDA approved for treatment of advanced cancer of the colon or rectum. The drugs are not approved for small bowel or ampulla of Vater cancer. Their use together in this study is investigational. Up to 30 people will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the small bowel or ampulla of Vater that is either unresectable or metastatic.
2. Patients must have measurable disease as per the modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
3. Patients may be previously untreated or have received previous systemic therapy, limited to 5-FU/leucovorin or capecitabine, as adjuvant or neoadjuvant therapy or as a radiosensitizer. Patients may have received capecitabine or 5-FU administered as a radiosensitizing agent concurrently with external beam radiotherapy as preoperative or postoperative therapy. Patients may have received capecitabine or 5-FU/leucovorin as part of adjuvant chemotherapy.
4. If radiation was previously received, the measurable disease must be outside the previous radiation field.
5. A minimum of 4 weeks must have elapsed since completion of any prior chemotherapy or radiotherapy. A minimum of 4 weeks must have elapsed since any prior surgery.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of less than or equal to 2.
7. Adequate bone marrow function defined as absolute peripheral granulocyte count of greater than or equal to 1500 mm3, platelet count greater than or equal to 1500 mm3, and hemoglobin greater than or equal to 10 gm/dL.
8. Adequate renal function, defined as serum creatinine less than or equal to 1.5 * ULN and calculated creatinine clearance >30 mL/min.
9. Patients must have adequate hepatic function: total bilirubin less than or equal to 1.5 gm/dL; serum albumin greater than or equal to 2.5 gm/dL. If the patient does not have liver metastasis, transaminases may be up to 2 * the ULN. If the patient has liver metastasis, transaminases up to 5 * Upper Limit of Normal (ULN) are allowed.
10. Negative urine or serum pregnancy test in women with childbearing potential, within one week prior to initiation of treatment.
11. The effects of the combination of oxaliplatin and capecitabine on the developing fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately.
12. Patients must sign an Informed Consent and Authorization indicating that they are aware of the investigational nature of this study and the known risks involved.
13. Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of XELOX in patients <18 years of age, children are excluded from this study.
14. Patients taking therapeutic doses of coumarin-derivative anticoagulants should be switched to low-molecular-weight heparin (LMWH). Low-dose Coumadin (e.g. 1 mg by mouth (PO) per day) in patients with in-dwelling venous access devices is allowed.

Exclusion Criteria:

1. Patients with prior exposure to platinum therapy are excluded. Patients who have received prior chemotherapy for metastatic disease are excluded.
2. Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or Mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
3. Patients may not be receiving any other investigational agents nor have received any investigational drug 30 days prior to enrollment.
4. Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and their risk for progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
5. Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation. Prior surgical therapy affecting absorption.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with XELOX. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
8. Patients with extensive symptomatic fibrosis of the lungs.
9. Peripheral neuropathy > grade 1.
10. Known Dihydropyrimidine dehydrogenase deficiency (DPD deficiency)
11. Patients receiving therapeutic doses of coumarin-derivative anticoagulant therapy are excluded since a drug interaction between capecitabine and coumarin anticoagulants has been reported. Patients requiring anticoagulation who may be safely switched to LMWH are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Wolff, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Overman MJ, Varadhachary GR, Kopetz S, Adinin R, Lin E, Morris JS, Eng C, Abbruzzese JL, Wolff RA. Phase II study of capecitabine and oxaliplatin for advanced adenocarcinoma of the small bowel and ampulla of Vater. J Clin Oncol. 2009 Jun 1;27(16):2598-603. doi: 10.1200/JCO.2008.19.7145. Epub 2009 Jan 21. PMID 19164203
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 1, 2004 and July 31, 2007. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Thirty-one patients were enrolled onto the study, and 30 patients received study treatment. One patient did not meet eligibility criteria and did not receive any study treatment. One additional patient was removed from the study after one treatment cycle.
Period: Overall Study
Arm/Group | Oxaliplatin + Capecitabine
Started | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin + Capecitabine
Number analyzed (Participants) | 30
Age Continuous [Median (Full Range); unit: years] | 62 [41 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Overall response rate defined as Complete Response (CR), disappearance of all target lesions; or Partial Response (PR), at least a 30% decrease in sum of longest diameter (LD) of target lesions, taking as reference the baseline sum LD, assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000]. In addition to a baseline scan, confirmatory scans for those deemed to have achieved a PR or CR.
Time Frame: Every 9 weeks from treatment initiation and confirmatory images 6 weeks or more after initial responses
Population: Analysis was intent-to-treat; One patient developed an acute flare of Crohn's disease after one cycle of study treatment and was removed from study without undergoing restaging scans.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin + Capecitabine
Number analyzed (Participants) | 30
participants
  Participants with CR | 3
  Participants with PR | 12

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from November 18, 2004 to July 26, 2007 or a total of three (3) years and five (5) months.
Arm/Group | Oxaliplatin + Capecitabine
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 30/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin + Capecitabine (N=30)
Abdominal Pain (Gastrointestinal disorders) | 12
Abdominal bloating (Gastrointestinal disorders) | 3
Alkaline Phosphatase (Metabolism and nutrition disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 6
Anorexia (Gastrointestinal disorders) | 17
Belching (Gastrointestinal disorders) | 2
Bilirubin (Metabolism and nutrition disorders) | 4
Chest Pain (Cardiac disorders) | 2
Cold Intolerance (General disorders) | 2
Constipation (Gastrointestinal disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 2
Decreased Total Protein, Serum (Metabolism and nutrition disorders) | 2
Dehydration (General disorders) | 3
Diarrhea (Gastrointestinal disorders) | 19
Dizziness (General disorders) | 6
Dry Eyes (Eye disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 5
Dry mouth (General disorders) | 4
Dysphagia (General disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Edema (limb) (Vascular disorders) | 6
Elevated phosphorus (Metabolism and nutrition disorders) | 2
Fatigue (General disorders) | 22
Fever without neutropenia (General disorders) | 9
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 6
Headache (General disorders) | 11
Heartburn (General disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 8
Hemorrhage (abdominal wound) (Gastrointestinal disorders) | 2
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypoatremia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Infection without neutropenia (Infections and infestations) | 3
Insomnia (General disorders) | 2
Irregular Menses (Reproductive system and breast disorders) | 2
Mood alteration(depression) (General disorders) | 11
Mucositis (Oral Cavity) (General disorders) | 6
Nausea (Gastrointestinal disorders) | 25
Neuropathy-Sensory (General disorders) | 28
Neutophils/granulocytes(ANC/AGC) (Blood and lymphatic system disorders) | 12
Pain (Muscle) (General disorders) | 14
Pain(joint) (Musculoskeletal and connective tissue disorders) | 12
Pain(throat/larynx) (General disorders) | 2
Platelets decreased (Metabolism and nutrition disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash desquamation (Skin and subcutaneous tissue disorders) | 9
Rash(hand/foot skin reaction) (Skin and subcutaneous tissue disorders) | 4
Rigors (Chills) (General disorders) | 8
Serum Glutamic Oxaloacetic Transaminase (AST,SGOT) (Metabolism and nutrition disorders) | 22
Serum Glutamic Pyruvic Transaminase (ALT,SGPT) (Metabolism and nutrition disorders) | 12
Taste Alteration (General disorders) | 9
Total elevated protein (Metabolism and nutrition disorders) | 4
Urinary Tract Infection (Renal and urinary disorders) | 3
Vomiting (Gastrointestinal disorders) | 19
Watery Eyes (Eye disorders) | 6
Weight Loss (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No